CLINICAL TRIAL: NCT04983901
Title: An Investigator Initiated, Phase II Single-Center, Randomized, Open-Label, Prospective, Study To Determine The Impact Of Serial Procalcitonin On Improving Antimicrobial Stewardship And On The Efficacy, Safety, And Tolerability Of Imipenem-Cilastatin-Relebactam Plus/Minus Vancomycin Or Linezolid Versus Standard Of Care Antipseudomonal Beta-Lactams Plus/Minus Vancomycin Or Linezolid As Empiric Therapy In Febrile Neutropenic Adults With Cancer
Brief Title: PHASE II SINGLE-CENTER, RANDOMIZED, OPEN-LABEL, PROSPECTIVE, STUDY TO DETERMINE THE IMPACT OF SERIAL PROCALCITONIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0074; NCI-2021-01957 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0074 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-07

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — imipenem, cilastatin and relebactam; Cefepime; Meropenem; Piperacillin, Tazobactam Drug Combination; Vancomycin; Daptomycin; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (imipenem, cilastatin, relebactam) (Experimental): Patients receive imipenem/cilastatin/relebactam IV over 30-60 minutes q6h for 2 days for a minimum of 8 doses. Patients may also receive gram-positive therapy at the discretion of the primary team or emergency center physician consisting of vancomycin IV q12h or linezolid IV or PO q12h. Patients may continue to receive imipenem/cilastatin/relebactam IVover 30-60 minutes for up to 14 days if clinically indicated by the assessment of the treating physician.
  Interventions: Drug: Imipenem/Cilastatin/Relebactam; Drug: Vancomycin; Drug: Daptomycin; Drug: Linezolid
- Group II (cefepime, meropenem, piperacillin/tazobactam) (Active Comparator): Patients receive cefepime IV q8h for a minimum of 6 doses, meropenem IV q8h for a minimum of 6 doses, or piperacillin/tazobactam IV q6h for a minimum of 8 doses. Patients may also receive gram-positive therapy at the discretion of the primary team or emergency center physician consisting of vancomycin IV q12h or linezolid IV or PO q12h.
  Interventions: Drug: Cefepime; Drug: Meropenem; Drug: Piperacillin-Tazobactam; Drug: Vancomycin; Drug: Daptomycin; Drug: Linezolid

INTERVENTIONS:
Drug: Imipenem/Cilastatin/Relebactam — Given IV
  Other Names: RECARBRIO™
  Arms: Group I (imipenem, cilastatin, relebactam)
Drug: Cefepime — Given IV
  Arms: Group II (cefepime, meropenem, piperacillin/tazobactam)
Drug: Meropenem — Given IV
  Other Names: Meropenem Trihydrate; Merrem I.V.; SM-7338
  Arms: Group II (cefepime, meropenem, piperacillin/tazobactam)
Drug: Piperacillin-Tazobactam — Given IV
  Other Names: PIPER/TAZO; Piperacillin/Tazobactam; Zosyn
  Arms: Group II (cefepime, meropenem, piperacillin/tazobactam)
Drug: Vancomycin — Given IV
Drug: Daptomycin — Given IV
  Other Names: Cubicin; LY146032
Drug: Linezolid — Given IV or PO
  Other Names: Zyvox

SUMMARY:
This phase II trial studies the effect of imipenem-relebactam in treating patients with cancer who have a fever due to low white blood cell counts (febrile neutropenia). In this study, imipenem-relebactam will be compared to the standard-of-care treatment (cefepime, meropenem, or piperacillin/tazobactam) for the treatment of febrile neutropenia. Imipenem-relebactam is used to treat infections. Giving imipenem-relebactam may help to control febrile neutropenia in patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of imipenem-relebactam plus vancomycin, daptomycin, or linezolid compared with SOC plus vancomycin, daptomycin or linezolid as empiric therapy in febrile neutropenic adults with cancer.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (TREATMENT): Patients receive imipenem/cilastatin/relebactam IV over 30-60 minutes once every 6 hours (q6h) for 2 days for a minimum of 8 doses. Patients may also receive gram-positive therapy at the discretion of the primary team or emergency center physician consisting of vancomycin IV q12h or linezolid IV or orally (PO) q12h. Patients may continue to receive imipenem/cilastatin/relebactam IV over 30-60 minutes for up to 14 days if clinically indicated by the assessment of the treating physician.

GROUP II (STANDARD OF CARE): Patients receive cefepime IV q8h for a minimum of 6 doses, meropenem IV q8h for a minimum of 6 doses, or piperacillin/tazobactam IV q6h for a minimum of 8 doses. Patients may also receive gram-positive therapy at the discretion of the primary team or emergency center physician consisting of vancomycin IV q12h or linezolid IV or PO q12h.

Patients in both groups may receive other additional therapy (double-gram negative therapy) consisting of tobramycin IV q24h, amikacin IV q24h, ciprofloxacin IV q8h, minocycline q12h, tigecycline on days 1-2 q12h, doxycycline q12h, and/or bactrim. After at least 48 hours of gram-negative antimicrobial therapy, patients may be allowed to switch to PO or IV therapy such as linezolid PO, ampicillin, amoxicillin, amoxicillin/clavulanate PO, minocycline PO, ciprofloxacin PO, levofloxacin PO, cefpodoxime PO, trimethoprim/sulfamethoxazole PO, ceftriaxone IV, ertapenem IV, daptomycin IV and/or vancomycin IV for outpatient or home administration as clinically indicated. While in the hospital, patients undergo the collection of blood samples daily for 2 weeks, and urine samples every 2 days for up to 2 weeks.

After completion of study treatment, patients are followed up at 2, 21-28, and 35-42 days.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent, and has the willingness and ability to comply with all study procedures
* >= 18 years old
* Patients with neutropenic fever who have existing malignancy or have undergone hematopoietic stem cell transplantation
* Neutropenic fever is defined as the presence of neutropenia defined by:

  * Absolute neutrophil count (ANC) < 500 cells/mm3 or has an ANC that is expected to decrease to < 500 cells/mm^3 within 48 hours of trial entry and fever defined as:
* Single oral temperature measurement of > 100.4 degree F (38.0 degree C).
* Requires hospitalization for IV empiric antibiotic therapy
* If female:

  * Not breastfeeding
  * Agrees to not attempt to become pregnant during the study. Is surgically sterile or at least 2-years postmenopausal, or if of childbearing potential, has negative screening serum or urine pregnancy test within 5 days
  * If of childbearing potential (including being < 2 years postmenopausal), is willing to practice sexual abstinence or use an effective dual form of contraception with her partner (eg, 2 barrier methods, barrier method plus hormonal method) during treatment and up 28 days post treatment

Exclusion Criteria:

* History of any hypersensitivity or allergic reaction to any carbapenem
* Fever suspected to be caused by a noninfectious cause (eg, fever related to drug or blood product administration)
* Confirmed fungal infection (eg, Pneumocystis jirovecii etiology in patients with pneumonia) that justifies adding additional empiric antimicrobial therapy (eg, antifungals)
* Confirmed viral infection that justifies adding additional empiric antiviral therapy (eg, ganciclovir, foscarnet)
* Evidence of significant hepatic impairment (any of the following):

  * Known acute viral hepatitis
  * Alanine aminotransferase (ALT) level > 5 times the upper limit of normal (x upper limit of normal [ULN]). Total bilirubin > 3 x ULN unless isolated hyperbilirubinemia is directly related to the acute infection or due to known Gilbert disease
  * Manifestations of end-stage liver disease, such as ascites or hepatic encephalopathy
* Known to be human immunodeficiency virus positive
* Severely impaired renal function, defined as creatinine clearance (CrCl) =< 30 mL/min estimated by the Cockcroft-Gault formula
* Expected requirement for hemodialysis while on study therapy
* Received > 36 hours of IV antibacterial therapy (with study drugs) within 72 hours of the initiation of inpatient IV study drug for treatment of suspected infection. Antibiotic prophylaxis and oral antibiotics is allowed. Prophylactic use of antiviral or antifungal medication is permitted
* Past or current history of epilepsy or seizure disorder; exception: well-documented febrile seizure of childhood
* Evidence of immediately life-threatening disease, progressively fatal disease, or life expectancy of 3 months or less (eg, moribund or with shock unresponsive to fluid replacement)
* Unable or unwilling to adhere to the study-specified procedures and restrictions
* Any condition that would make the patient, in the opinion of the Investigator, unsuitable for the study (eg, would place a patient at risk or compromise the quality of the data
* Participation in any other ongoing imipenem-relebactam trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam I Raad, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Dagher H, Chaftari AM, Hachem R, Jiang Y, Philip A, Mulanovich P, Haddad A, Lamie P, Wilson Dib R, John TM, Dailey Garnes NJM, Ali S, Chaftari P, Raad II. Procalcitonin Level Monitoring in Antibiotic De-Escalation and Stewardship Program for Patients with Cancer and Febrile Neutropenia. Cancers (Basel). 2024 Oct 11;16(20):3450. doi: 10.3390/cancers16203450. PMID 39456544
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 14, 2021 and October 06, 2023, patients presenting to the emergency medicine department were screened through an EPIC generated list identifying patients with fever and neutropenia that meet the inclusion criteria.
Groups:
- Imipenem-Relebactam Arm: Patients receive imipenem/cilastatin/relebactam IV over 30-60 minutes once every 6 hours (q6h) for 2 days for a minimum of 8 doses. May also receive gram-positive therapy consisting of vancomycin IV q 12h or linezolid IV or orally (PO) q12h. Daptomycion could be given if no pneumonia. Participants may continue on the study drug for up to 14 days. Participants may receive other addtional therapy.
- Standard of Care (SOC) Arm: Patients receive cefepime IV q8h for a minimum of 6 doses, or meropenem IV q8h for a minimum of 6 doses, or piperacillin/tazobactam IV q6h for a minimum of 8 doses. May also receive gram-positive therapy consisting of vancomycin IV q 12h or linezolid IV or orally (PO) q12h. Daptomycion could be given if no pneumonia. Patients may receive other additional therapy.
Period: Overall Study
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Started | 50 | 50
Completed | 44 | 44
Not Completed | 6 | 6
Not completed — Death | 1 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Patients in Modified Intent-To-Treat (MITT) analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Median (Full Range); unit: years] | 55 [18 to 80] | 63 [21 to 84] | 61 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 26 | 27 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 1 | 4
  Black or African American | 4 | 5 | 9
  Hispanic or Latino | 8 | 4 | 12
  Middle East | 1 | 1 | 2
  White | 33 | 38 | 71
  Others | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99
Type of Cancer [Count of Participants; unit: Participants]
  Hematological malignancy | 33 | 31 | 64
  Solid tumor | 16 | 19 | 35
History of BMT within one year [Count of Participants; unit: Participants] — Population: History of BMT within one year
  Participants
    History of BMT within one year | 3 | 6 | 9
    Autologous | 0 | 3 | 3
    Allogeniec | 3 | 3 | 6
Type of allogeneic transplant [Count of Participants; unit: Participants]
  Matched unrelated donor | 2 | 2 | 4
  HLA matched related | 1 | 0 | 1
  Others | 0 | 1 | 1
  GVHD | 2 | 2 | 4
Temperature at initial presentation (oC) [Count of Participants; unit: Participants]
  < 36 | 0 | 0 | 0
  36-38 | 0 | 0 | 0
  > 38 | 49 | 50 | 99
Sepsis status [Count of Participants; unit: Participants]
  No sepsis | 35 | 35 | 70
  Sepsis | 14 | 14 | 28
  Severe sepsis | 0 | 1 | 1
Neurologic impairment [Count of Participants; unit: Participants]
  Neurologic impairment | 1 | 0 | 1
  Confusion | 1 | 0 | 1
Clinical source presentation [Count of Participants; unit: Participants] | 26 | 25 | 51
Site of clinical presentation [Count of Participants; unit: Participants]
  Head and neck | 1 | 0 | 1
  Lung (pneumonia) | 18 | 19 | 37
  Abdomen | 7 | 4 | 11
  Genitourinary | 1 | 2 | 3
  Skin and soft tissue | 1 | 1 | 2
Microbiological documentation (positivity) [Count of Participants; unit: Participants] | 13 | 17 | 30
Site of organism [Count of Participants; unit: Participants]
  Genitourinary | 0 | 2 | 2
  Blood | 13 | 15 | 28
Organisms identified [Count of Participants; unit: Participants]
  Organisms identified | 13 | 17 | 30
  Gram negative | 7 | 8 | 15
  Gram positive | 6 | 5 | 11
  Both Gram Positive and Gram Negative | 0 | 4 | 4
Organisms recovered in positive cultures [Count of Participants; unit: Participants]
  Organisms recovered in positive cultures | 13 | 17 | 30
  Enterobacter cloacae | 2 | 1 | 3
  Escherichia coli | 3 | 3 | 6
  Klebsiella pneumoniae | 0 | 2 | 2
  Pseudomonas aeruginosa | 1 | 2 | 3
  Rhizobium radiobacter | 1 | 0 | 1
  Klebsiella pneumoniae & Enterococcus faecalis | 0 | 1 | 1
  Haemophilus parainfluenzae & Streptococcus mitis/oralis Group | 0 | 1 | 1
  Pseudomonas aeruginosa, Streptococcus mitis/oralis Group & Enterococcus faecalis | 0 | 1 | 1
  Roseomonas mucosa, Micrococcus luteus & Dermacoccus nishinomiyaensis | 0 | 1 | 1
  Enterococcus faecium | 0 | 1 | 1
  Staphylococcus epidermidis | 1 | 2 | 3
  Streptococcus mitis/oralis group | 4 | 2 | 6
  Enterococcus faecalis & Rothia mucilaginosa | 1 | 0 | 1
Bacteremia [Count of Participants; unit: Participants] | 13 | 15 | 28
CVC being the source of BSI isolation [Count of Participants; unit: Participants] | 12 | 11 | 23
SOC Antibiotics [Count of Participants; unit: Participants]
  Cefepime | 0 | 43 | 43
  Meropenem | 0 | 2 | 2
  Piperacillin/tazobactam | 0 | 5 | 5
Antibiotics for gram positive coverage [Count of Participants; unit: Participants]
  Vancomycin | 20 | 20 | 40
  Linezolid | 18 | 27 | 45
  Daptomycin | 3 | 1 | 4
  Linezolid & daptomycin | 1 | 0 | 1
  None | 7 | 2 | 9
Gram positive coverage with any of the above antibiotics [Count of Participants; unit: Participants] | 42 | 48 | 90
ICU admission [Count of Participants; unit: Participants] | 3 | 2 | 5
Mechanical ventilation [Count of Participants; unit: Participants] | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcome in the MITT Analysis Set at EOIV.
Description: The primary efficacy outcome is favorable clinical response of the patients in the MITT (Modified Intent-To-Treat) Analysis Set at end of inpatient intravenous therapy (EOIV). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug.
Population: Patients in MITT (Modified Intent-To-Treat) Analysis Set The MITT Analysis Set will be a subset of the ITT Analysis Set and will include all randomized patients who received any amount of inpatient IV study drug and meet minimal disease criteria (Inclusion Criterion 3). Patients will be analyzed according to randomized treatment group, regardless of treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 49 | 50
Participants
  Favorable clinical resposne | 44 | 37
  Clinical failure | 5 | 12
  Indeterminate | 0 | 1

2. Secondary Outcome: Clinical Outcome in the mMITT Analysis Set at EOIV.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at end of inpatient intravenous therapy (EOIV). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug.
Population: Patients in mMITT (Microbiological Modified Intent-To-Treat) Analysis Set The mMITT Analysis Set will be a subset of the MITT Analysis Set and will include those patients for whom at least 1 qualifying bacterial pathogen was isolated from an appropriate microbiological specimen at baseline, irrespective of susceptibility to study therapies
Measure: Count of Participants; unit: Participants
Groups:
- Imipenem-Relebactam Arm: Patients receive imipenem/cilastatin/relebactam IV over 30-60 minutes once every 6 hours (q6h) for 2 days for a minimum of 8 doses. May also receive gram-positive therapy consisting of vancomycin IV q 12h or linezolid IV or orally (PO) q12h. Daptomycion could be given if no pneumonia. Participants may continue on the study drug for up to 14 days. Patients may receive other addtional therapy.
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 7 | 12
Participants
  Favorable clinical resposne | 6 | 8
  Clinical failure | 1 | 3
  Indeterminate | 0 | 1

3. Secondary Outcome: Clinical Outcome in the CE Analysis Set at EOIV.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the CE (Clinically Evaluable) Analysis Set at end of inpatient intravenous therapy (EOIV). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug.
Population: Patients in CE (Clinically Evaluable) Analysis Set - A subset of the MITT Analysis Set including patients with the following conditions:
  Received >=48 hrs of IV study drug to be considered an evaluable clinical failure, unless deemed a clinical failure based on a treatment-limiting AE Received >=48 hrs of IV gram negative coverage to be considered an evaluable clinical cure Had clinical outcome assessment at TOC (other than indeterminate) or assessed as clinical failure at EOIV or TOC
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 42 | 35
Participants
  Favorable clinical resposne | 37 | 26
  Clinical failure | 5 | 9

4. Secondary Outcome: Clinical Outcome in the MITT Analysis Set at TOC.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the MITT (Modified Intent-To-Treat) Analysis Set at test-of-cure (TOC). The clinical outcome has three categories: Clinical cure, Clinical failure, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug.
Population: Pateints in MITT (Modified Intent-To-Treat) Analysis Set The MITT Analysis Set will be a subset of the ITT Analysis Set and will include all randomized patients who received any amount of inpatient IV study drug and meet minimal disease criteria (Inclusion Criterion 3). Patients will be analyzed according to randomized treatment group, regardless of treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 49 | 50
Participants
  Clinical cure | 35 | 32
  Clinical failure | 8 | 13
  Indeterminate | 6 | 5

5. Secondary Outcome: Clinical Outcome in the MITT Analysis Set at LFU.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the MITT (Modified Intent-To-Treat) Analysis Set at late follow-up (LFU). The clinical outcome has three categories: Clinical cure, Clinical failure, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Imipenem-Relebactam Arm: Patients receive imipenem/cilastatin/relebactam IV over 30-60 minutes once every 6 hours (q6h) for 2 days for a minimum of 8 doses. May also receive gram-positive therapy consisting of vancomycin IV q 12h or linezolid IV or orally (PO) q12h. Daptomycion could be given if no pneumonia. Participants may continue on the study drug for up to 14 days. Patients may receive other additional therapy.
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 49 | 50
Participants
  Clinical cure | 33 | 30
  Clinical failure | 8 | 13
  Indeterminate | 8 | 7

6. Secondary Outcome: Clinical Outcome in the mMITT Analysis Set at TOC.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at test-of-cure (TOC). The clinical outcome has three categories: Clinical cure, Clinical failure, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 7 | 12
Participants
  Clinical cure | 3 | 6
  Clinical failure | 2 | 4
  Indeterminate | 2 | 2

7. Secondary Outcome: Clinical Outcome in the mMITT Analysis Set at LFU.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at late follow-up (LFU). The clinical outcome has three categories: Clinical cure, Clinical failure, and Indeterminate.
Time Frame: Pateints in mMITT (Microbiological Modified Intent-To-Treat) Analysis Set
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 7 | 12
Participants
  Clinical cure | 3 | 6
  Clinical failure | 2 | 4
  Indeterminate | 2 | 2

8. Secondary Outcome: Clinical Outcome in the CE Analysis Set at TOC.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the CE (Clinically Evaluable) Analysis Set at test-of-cure (TOC). The clinical outcome has three categories: Clinical cure, Clinical failure, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 42 | 35
Participants
  Clinical cure | 34 | 25
  Clinical failure | 8 | 10

9. Secondary Outcome: Clinical Outcome in the CE Analysis Set at LFU.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the CE (Clinically Evaluable) Analysis Set at late follow-up (LFU). The clinical outcome has three categories: Clinical cure, Clinical failure, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Imipenem-Relebactam Arm: Patients receive imipenem/cilastatin/relebactam IV over 30-60 minutes once every 6 hours (q6h) for 2 days for a minimum of 8 doses. May also receive gram-positive therapy consisting of vancomycin IV q 12h or linezolid IV or orally (PO) q12h. Daptomycion could be given if no pneumonia. Patients may continue on the study drug for up to 14 days. Patients may receive other addtional therapy.
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 42 | 35
Participants
  Clinical cure | 32 | 23
  Clinical failure | 8 | 10
  Indeterminate | 2 | 2

10. Secondary Outcome: Clinical Outcome in the ME Analysis Set at EOIV.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the ME (Microbiologically Evaluable) Analysis Set at end of inpatient intravenous therapy (EOIV). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug.
Population: Patients in ME (Microbiologically Evaluable) Analysis Set The ME Analysis Set will include patients who meet the criteria for both the CE and mMITT analysis sets.
Measure: Count of Participants; unit: Participants
Groups:
- Imipenem-Relebactam Arm: Patients receive imipenem/cilastatin/relebactam IV over 30-60 minutes once every 6 hours (q6h) for 2 days for a minimum of 8 doses. May also receive gram-positive therapy consisting of vancomycin IV q 12h or linezolid IV or Patients may continue on the study drug for up to 14 days. Patients may receive other addtional therapy.
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 5 | 7
Participants
  Favorable clinical resposne | 4 | 6
  Clinical failure | 1 | 1

11. Secondary Outcome: Clinical Outcome in the ME Analysis Set at TOC.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the ME (Microbiologically Evaluable) Analysis Set at test-of-cure (TOC). The clinical outcome has three categories: Clinical cure, Clinical failure, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Groups:
- Imipenem-Relebactam Arm: Patients receive imipenem/cilastatin/relebactam IV over 30-60 minutes once every 6 hours (q6h) for 2 days for a minimum of 8 doses. May also receive gram-positive therapy consisting of vancomycin IV q 12h or linezolid IV or Patients may continue on the study drug for up to 14 days. Patients may receive other additional therapy.
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 5 | 7
Participants
  Clinical cure | 3 | 5
  Clinical failure | 2 | 2

12. Secondary Outcome: Clinical Outcome in the ME Analysis Set at LFU.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the ME (Microbiologically Evaluable) Analysis Set at late follow-up (LFU). The clinical outcome has three categories: Clinical cure, Clinical failure, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 5 | 7
Participants
  Clinical cure | 3 | 5
  Clinical failure | 2 | 2

13. Secondary Outcome: Microbiological Outcome in the mMITT Analysis Set at EOIV.
Description: The secondary efficacy outcome is favorable microbiological response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at end of inpatient intravenous therapy (EOIV). The microbiological response outcome has five categories: Persistence, eradication, presumed eradication, presumed persistence, and Indeterminate.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 7 | 12
Participants
  Eradication | 7 | 9
  Presumed eradication | 0 | 2
  Indeterminate | 0 | 1

14. Secondary Outcome: Microbiological Outcome in the mMITT Analysis Set at TOC.
Description: The secondary efficacy outcome is favorable microbiological response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at test-of-cure (TOC). The microbiological response outcome has five categories: Persistence, eradication, presumed eradication, presumed persistence, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 7 | 12
Participants
  Eradication | 5 | 10
  Presumed eradication | 0 | 1
  Indeterminate | 2 | 1

15. Secondary Outcome: Microbiological Outcome in the mMITT Analysis Set at LFU.
Description: The secondary efficacy outcome is favorable microbiological response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at late follow-up (LFU). The microbiological response outcome has five categories: Persistence, eradication, presumed eradication, presumed persistence, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 7 | 12
Participants
  Eradication | 5 | 10
  Presumed eradication | 0 | 1
  Indeterminate | 2 | 1

16. Secondary Outcome: Microbiological Outcome in the ME Analysis Set at EOIV.
Description: The secondary efficacy outcome is favorable microbiological response of the patients in the ME (Microbiologically Evaluable) Analysis Set at end of inpatient intravenous therapy (EOIV). The microbiological response outcome has five categories: Persistence, eradication, presumed eradication, presumed persistence, and Indeterminate.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 5 | 7
Participants
  Eradication | 5 | 5
  Presumed eradication | 0 | 2

17. Secondary Outcome: Microbiological Outcome in the ME Analysis Set at TOC.
Description: The secondary efficacy outcome is favorable microbiological response of the patients in the ME (Microbiologically Evaluable) Analysis Set at test-of-cure (TOC). The microbiological response outcome has five categories: Persistence, eradication, presumed eradication, presumed persistence, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 5 | 7
Participants
  Eradication | 5 | 6
  Presumed eradication | 0 | 1

18. Secondary Outcome: Microbiological Outcome in the ME Analysis Set at LFU.
Description: The secondary efficacy outcome is favorable microbiological response of the participants in the ME (Microbiologically Evaluable) Analysis Set at late follow-up (LFU). The microbiological response outcome has five categories: Persistence, eradication, presumed eradication, presumed persistence, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 5 | 7
Participants
  Eradication | 5 | 6
  Presumed eradication | 0 | 1

19. Secondary Outcome: Infection-related Mortality in the MITT Analysis Set at TOC.
Description: The secondary efficacy outcome is infection-related mortality of the patients in the MITT (Modified Intent-To-Treat) Analysis Set at test-of-cure (TOC).
Time Frame: 21 to 28 days after the start of inpatient IV study drug.
Population: Participants in MITT (Modified Intent-To-Treat) Analysis Set The MITT Analysis Set will be a subset of the ITT Analysis Set and will include all randomized patients who received any amount of inpatient IV study drug and meet minimal disease criteria (Inclusion Criterion 3). Patients will be analyzed according to randomized treatment group, regardless of treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 49 | 50
Participants | 0 | 0

20. Secondary Outcome: Infection-related Mortality in the MITT Analysis Set at LFU.
Description: The secondary efficacy outcome is infection-related mortality of the patients in the MITT (Modified Intent-To-Treat) Analysis Set at late follow-up (LFU).
Time Frame: 35 to 42 days after the start of inpatient IV study drug.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 49 | 50
Participants | 0 | 0

21. Secondary Outcome: Infection-related Mortality in the mMITT Analysis Set at TOC.
Description: The secondary efficacy outcome is Infection-related mortality of the participants in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at test-of-cure (TOC).
Time Frame: 21 to 28 days after the start of inpatient IV study drug.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care (SOC) Arm: Participants receive cefepime IV q8h for a minimum of 6 doses, or meropenem IV q8h for a minimum of 6 doses, or piperacillin/tazobactam IV q6h for a minimum of 8 doses. May also receive gram-positive therapy consisting of vancomycin IV q 12h or linezolid IV or orally (PO) q12h. Daptomycion could be given if no pneumonia. Participants may receive other additional therapy.
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 7 | 12
Participants | 0 | 0

22. Secondary Outcome: Infection-related Mortality in the mMITT Analysis Set at LFU.
Description: The secondary efficacy outcome is Infection-related mortality of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at late follow-up (LFU).
Time Frame: 35 to 42 days after the start of inpatient IV study drug.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 7 | 12
Participants | 0 | 0

23. Secondary Outcome: 30-Day All-cause Mortality in the MITT Analysis Set.
Description: The secondary efficacy outcome is 30-day all-cause mortality of the patients in the MITT (Modified Intent-To-Treat) Analysis Set.
Time Frame: 30 days after the last dose of inpatient IV study drug.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 49 | 50
Participants | 2 | 3

24. Secondary Outcome: 30-Day All-cause Mortality in the mMITT Analysis Set.
Description: The secondary efficacy outcome is 30-day all-cause mortality of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set.
Time Frame: 30 days after the last dose of inpatient IV study drug.
Population: Patients in MITT (Modified Intent-To-Treat) Analysis Set The mMITT Analysis Set will be a subset of the MITT Analysis Set and will include those patients for whom at least 1 qualifying bacterial pathogen was isolated from an appropriate microbiological specimen at baseline, irrespective of susceptibility to study therapies.
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem-Relebactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 7 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of the start of inpatient IV study drug to 35 to 42 days after the start of inpatient IV study drug
Description: Per protocol, all SAEs were collected and reported according to the clinicaltrials.gov definitions.
  Per protocol, all AEs of any grade that are possibly, probably and definitely related to the study drug, and any AE grade 3 or above regardless of their attribution to study drug were collected and reported. Therefore, other AEs, not required per protocol, were not collected.
Groups:
- Group II (Cefepime, Meropenem, Piperacillin/Tazobactam): Patients receive cefepime IV q8h for a minimum of 6 doses, or meropenem IV q8h for a minimum of 6 doses, or piperacillin/tazobactam IV q6h for a minimum of 8 doses. May also receive gram-positive therapy consisting of vancomycin IV q 12h or linezolid IV or orally (PO) q12h. Daptomycion could be given if no pneumonia. Patients may receive other additional therapy.
Arm/Group | Imipenem-Relebactam Arm | Group II (Cefepime, Meropenem, Piperacillin/Tazobactam)
All-Cause Mortality (participants affected / at risk) | 1/49 | 4/50
Serious Adverse Events (participants affected / at risk) | 30/49 | 29/50
Other Adverse Events (participants affected / at risk) | 4/49 | 7/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imipenem-Relebactam Arm (N=49) | Group II (Cefepime, Meropenem, Piperacillin/Tazobactam) (N=50)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Blood and lymphatic system disorders - Other: Ileocolic lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 13 | 7
Atrial fibrillation (Cardiac disorders) | 1 | 0
Heart Failure (Cardiac disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic Obstruction (Gastrointestinal disorders) | 1 | 0
Gastric Hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other: enteritis (Gastrointestinal disorders) | 0 | 1
Jejunal perforation (Gastrointestinal disorders) | 1 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
Fever (General disorders) | 2 | 2
Mutli-organ failure (General disorders) | 0 | 1
Immune system disorders - Other: ICANS (Immune system disorders) | 1 | 0
Anorectal Infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 3
Catheter related bloodstream infection (Infections and infestations) | 2 | 1
Fungemia (Infections and infestations) | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 1
Infections and infestations others Hidradenitis of the Right Axilla (Infections and infestations) | 0 | 1
Infections and infestations, other specigy: COVID19 (Infections and infestations) | 0 | 1
Kidney Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 8 | 10
Salivary gland infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 8 | 2
Sinusitis (Infections and infestations) | 1 | 0
skin infection (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0
Soft Tissue Infection - Cellulitis (Infections and infestations) | 1 | 1
Upper Respiratory Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Injury To Carotid Artery (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 2
CPK increased (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intracranial Hemorrhage (Nervous system disorders) | 1 | 0
Nervous system disorders - Other: Ring-enhancing brain lesions (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Genital edema (Reproductive system and breast disorders) | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Reproductive system and breast disorders) | 1 | 3
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders Other, specify Chronic and Acute Skin Lesions (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial thromboembolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imipenem-Relebactam Arm (N=49) | Group II (Cefepime, Meropenem, Piperacillin/Tazobactam) (N=50)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Allergic Reaction (Immune system disorders) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 4
Aspartate Aminotransferase Increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
CPK increased (Investigations) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other red rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT04983901/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT04983901/ICF_001.pdf